CLINICAL TRIAL: NCT06276543
Title: A Multi-center, Retrospective Registry Study on the Safety of Bactiseal Catheter
Brief Title: Bactiseal Catheter Safety Registry Study
Status: Recruiting | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: C-BSEAL-002
Record Dates: First submitted 2024-02-08; First posted 2024-02-26 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Hydrocephalus
Keywords: hydrocephalus; cerebrospinal fluid; Shunt; antibiotic-impregnated catheter; infection
MeSH Terms: conditions — Hydrocephalus; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- antibiotic-impregnated catheter group: Hydrocephalus patients implanted with antibiotic-impregnated catheter.
  Interventions: Device: antibiotic-impregnated catheter

INTERVENTIONS:
Device: antibiotic-impregnated catheter — Hydrocephalus patient implant with antibiotic-impregnated catheter to shunt their cerebrospinal fluid.

SUMMARY:
Research Purpose:

This study aims to continuously evaluate the safety of subjects implanted with a catheter (trade name: Bactiseal) produced by Integra LifeSciences Production Corporation. Device safety will be assessed based on all the adverse events that occurred within 2 years after implanted the catheter.

Research Design:

This study is designed to be single arm, multi-center, and retrospective. A total of 200 subjects will be retrospectively enrolled. Information will be collected on adverse events, including bacterial culture and drug resistance testing when infection (if done), of subjects enrolled within 2 years after the implantation of the Bactiseal Catheter between January 01, 2019 and June 30, 2022.

The following information will be collected from subjects' medical records or hospitals' databases (if any):

1. General condition of the subjects (including previous shunting and external drainage operation)
2. Intraoperative condition and catheter implantation
3. Information on the shunt catheters
4. Adverse events of subjects within 2 years after the operation and classification of the adverse events (except anticipated adverse events listed in section 8.1.2)
5. Relevant examinations in case of postoperative infection, including bacterial culture and drug resistance testing (if done)

ELIGIBILITY:
Inclusion Criteria:

1. The informed consent is exempted by the Ethics Committee of a research center. Or a subject or his/her legal representative signed the informed consent form (ICF) prior to the enrollment.
2. A subject had an indication suitable to use Bactiseal Catheter.
3. A subject implanted hydrocephalus shunt catheter for at least 2 years at the time of enrollment.

Exclusion Criteria:

1. A subject didn't have an indication suitable to use the catheter.
2. A subject was known to be allergic to a component or ingredient of the catheter to be implanted, including silicone catheter, rifampicin, and clindamycin.
3. According to the comprehensive judgment of an investigator, a subject had an infection of the implant site when the shunt is implanted, such as ventriculitis, meningitis, peritonitis, and local implant skin infection.
4. A subject was simultaneously implanted with another shunt catheter different from Bactiseal Catheter.
5. A subject had a contraindication of the shunt operation.
6. A subject had uncorrected coagulopathy or any bleeding disorder.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 200 hydrocephalus patients will be enrolled and adverse events will be collected for those enrolled subjects within two years after the implantation of the Bactiseal catheter from January 01, 2019 to June 30, 2022, through reviewing subject record or hospital database.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09-29 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Infection outcome | 2 years post catheter implanted.
  Incidence of Bactiseal Shunt catheter related infection within 2 years post implant.
Safety outcome | 2 years post catheter implanted.
  Incidence of adverse events of a subject within 2 years post implant Bactiseal

CONTACTS AND LOCATIONS:
Overall Officials: Nan Bao, MD, Principal Investigator — Shanghai Children's Medical Center Affiliated to Shanghai Jiaotong University School of Medicine
Locations (8):
- China (8):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - the 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - the Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Shanghai Children's Medical Center affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No
individual participant data (IPD) is not available to other researchers.